CLINICAL TRIAL: NCT07232329
Title: Experimental and Quantitative Research Method
Brief Title: The Effect of Chronic Breathing Exercises on Pulmonary Functions: A Study on Combined Aerobic Exercise and Synchronized Breathing Exercises
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bandırma Onyedi Eylül University (Other)
Responsible Party: Principal Investigator, Ahmet KURTOĞLU, Assoc. Prof., Bandırma Onyedi Eylül University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-1
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2024-04

CONDITIONS: Pulmonary; Exercise; Breathing Exercise
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (Experimental)
  Interventions: Other: aerobic exercise with synchronized breathing group
- aerobic exercise group (Experimental)
  Interventions: Other: aerobic exercise with synchronized breathing group
- aerobic exercise with synchronized breathing group (Experimental)
  Interventions: Other: aerobic exercise with synchronized breathing group

INTERVENTIONS:
Other: aerobic exercise with synchronized breathing group — This study was ethically approved by the Bandirma Onyedi Eylül University Rectorate Health Sciences Non-Interventional Research Ethics Committee with the meeting decision numbered 2024-1 on 16.01.2024. Within the scope of the study, all participants were informed about the purpose of the study, the reason for the study, and its contribution to the literature. The participants were informed that this study would be conducted on a completely voluntary basis and that they could withdraw from the study at any time. This study was conducted in accordance with the principles set out in the Declaration of Helsinki. In this study, an experimental and quantitative research method including pre-test and post-test measurements will be used and the chronic effect of 8-week breathing exercises on pulmonary functions, heart rate, and peripheral oxygen saturation (SPO2) level will be examined. Participants' pulmonary function and resting heart rate will be measured

SUMMARY:
In this respect, the aim of this study was to investigate the effects of synchronous breathing exercise and aerobic exercise on pulmonary functions. In the study, three groups including a control group (CG), an aerobic exercise group (AE), and both breathing and aerobic exercise (AE+SB) were compared and analyzed. In the study, the accuracy of the following hypotheses was tried to be investigated. H1a "Synchronous breathing exercise has an impact on respiratory function." H1b "Aerobic exercises have an impact on respiratory function." H1c "Synchronized breathing exercises combined with aerobic exercises have a greater impact on respiratory function."

ELIGIBILITY:
Inclusion Criteria:

* healthy university students
* aged 18-25 years,
* sedentary lifestyle (150 min/week of physical activity)

Exclusion Criteria:

* history of cardiopulmonary disease,
* smoking,
* alcohol use,
* current infection,
* chronic medication use,
* recent hospitalization due to pulmonary conditions.
* involved in competitive sports.

Exclusion Criteria

- Participants not adhering to training sessions or instructions were also excluded.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Pre_Pulmonary Function Test | 8 weeks
Post_Pulmonary Function Test | 8 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Bandirma Onyedi Eylul University, Balıkesir, Bandırma
  - Sport Science Faculty Multiple Aimed Sport Hall, Balıkesir, Bandırma

IPD SHARING:
Plan to Share IPD: No
Participants have only been given permission for their data to be used within the scope of this research.